CLINICAL TRIAL: NCT01899742
Title: DB2116960: A Randomized, Double-Dummy, Parallel Group, Multicenter Trial Comparing the Efficacy and Safety of UMEC/VI (a Fixed Combination of Umeclidinium and Vilanterol) With Tiotropium In Subjects With COPD Who Continue To Have Symptoms on Tiotropium
Brief Title: The Purpose of the This Study is to Evaluate the Spirometric Effect (Trough FEV1) of Umeclidinium/Vilanterol 62.5/25 mcg Once Daily Compared With Tiotropium 18mcg Once Daily Over a a 12-week Treatment Period in Subjects With COPD Who Continue to Have Symptoms on Tiotropium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116960
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; vilanterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umeclidinium/Vilanterol (Experimental): Long-acting muscarinic antagonist (LAMA)/Long-acting Beta agonist (LABA)
  Interventions: Drug: Umeclidinium/Vilanterol 62.5/25 mcg
- Tiotropium (Active Comparator): Long-acting muscarinic antagonist (LAMA)
  Interventions: Drug: Tiotropium 18 mcg

INTERVENTIONS:
Drug: Umeclidinium/Vilanterol 62.5/25 mcg — Inhalation Powder
  Arms: Umeclidinium/Vilanterol
Drug: Tiotropium 18 mcg — Inhalation Powder
  Arms: Tiotropium

SUMMARY:
The primary objective is to compare the efficacy of UMEC/VI Inhalation Powder (62.5/25 mcg) once-daily with tiotropium (18 mcg) once-daily over 12 weeks for the treatment of subjects with COPD who have received tiotropium and continue to have symptoms while on tiotropium.

DETAILED DESCRIPTION:
This is a Phase IIIb multicentre, randomized, blinded, double-dummy, parallel group study to evaluate the efficacy and safety of UMEC/VI Inhalation Powder (62.5/25 mcg) when administered once-daily via ELLIPTA dry powder inhaler (DPI) [note: the ELLIPTA DPI may also be referred to as the Novel DPI (NDPI) or the DPI] compared with tiotropium (18 mcg) administered once-daily via the HandiHaler over a treatment period of 12 weeks in subjects with COPD who continue to have symptoms while on tiotropium.

The target population of the study will include those subjects who continue to have symptoms while on tiotropium. The study will screen approximately 650 subjects who continue to have symptoms whilst on tiotropium. After a 4 week run-in period on open label tiotropium, those subjects who continue to have symptoms and have adhered to the treatment schedule will progress into the treatment phase.

At the end of the run-in phase approximately 490 subjects will be randomised 1:1 to UMEC/VI Inhalation Powder (62.5/25 mcg), or tiotropium (18 mcg). During the treatment phase, each subject will receive two inhalers, a preloaded ELLIPTA DPI and a HandiHaler dry powder inhaler with capsules, for once-daily administration of one active treatment and one placebo treatment for 12 weeks.

There will be a total of 8 study visits. Subjects will sign the informed consent form (ICF) at either Visit 0 or Visit 1 and will be assigned a subject identifier. Subjects who meet the eligibility criteria at Screening (Visit 1) will enter the open label tiotropium run-in phase. After 4 weeks all subjects will be reviewed (Visit 2) and if they satisfy the randomisation criteria they will be randomised and enter the treatment phase.

After Visit 2, there will be a further 6 study clinic visits. Further visits are scheduled at Day 2, Week 4, Week 8, Week 12 and Week 12 +1 day (Visits 3 to 7 respectively). Vital signs (blood pressure and pulse rate) will be obtained at all clinic visits.

Trough FEV₁and trough FVC will be performed at Visit 3 and Visit 7. Pre-dose and post dose FEV₁and FVC measurement at 5 and 15 mins and 1 and 3 hrs will also be performed at Visit 2, Visit 4, Visit 5 and Visit 6.

At selected study sites, a subset of approximately 200 subjects will perform 24-hour serial spirometry at Visit 2 and Visit 6 for evaluation of lung function over the dosing period.

An assessment of dyspnea will be obtained using the Baseline and Transition Dyspnea Index (BDI/TDI). At Visit 2, the severity of dyspnea at baseline will be assessed using the BDI. Change from baseline will be assessed using the TDI at Visit 4, Visit 5 and Visit 6.

In addition to the baseline assessment at Visit 2, health status will be captured using the St. George Respiratory Questionnaire for COPD (SGRQ-C) scale at Visit 4 and Visit 6.

The impact of COPD on the subject's wellbeing and daily life will be measured using the COPD Assessment Test (CAT) and the the Euroqol-5D (EQ5D).. In addition to the baseline assessment at Visit 2, the CAT and the EQ-5D will also completed at Visit 4 and Visit 6. Furthermore, the CAT is also completed during screening.

The Patient Global Rating of COPD Severity and Change of COPD Severity is a selfreported global assessment of severity of illness will be performed at Baseline during Visit 2 and at Visit 4 and Visit 6.

Visits 0/1 through 7 will be clinic visits conducted on an outpatient basis. A safety Follow-Up assessment (Visit 8) will be conducted either by phone call or clinic visit where required approximately 7 days after the end of the study treatment (Visit 7 or Early Withdrawal, if applicable). The total duration of subject participation, including follow-up, will be approximately 18 weeks. All subjects will be provided with albuterol/salbutamol for use on an "as-needed" basis throughout the run-in and study treatment periods.

For determination of subject disposition, subjects will be considered to have completed the study upon completion of Visit 7 (the last on-treatment clinic visit). There are no plans for compassionate use of the study medications.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: Subjects 40 years of age or older at Visit 1.
* Gender: Male or female subjects. A female is eligible to enter and participate in the study if she is of:

Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, >45 years, in the absence of hormone replacement therapy.

OR

Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact):

* Abstinence
* Oral Contraceptive, either combined or progestogen alone
* Injectable progestogen
* Implants of levonorgestrel
* Estrogenic vaginal ring
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS) that meets the SOP effectiveness criteria as stated in the product label
* Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records.
* Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)

  * Bronchodilator Treatment: Subjects must have been prescribed tiotropium either via the HandiHaler device or Respimat for at least 3 months prior to screening (Visit 1).
  * COPD Diagnosis: A diagnosis of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society [Celli, 2004].
  * Smoking History: Current or former cigarette smokers with a history of cigarette smoking of ≥10 pack-years [number of pack years = (number of cigarettes per day /20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.

Note: Pipe and/or cigar use cannot be used to calculate pack-year history

* Severity of Disease: A pre and post-albuterol/salbutamol FEV₁/FVC ratio of <0.70 and post-albuterol/salbutamol FEV₁ of ≤70% and ≥50% predicted normal values calculated using reference equations at Visit 1 [Quanjer, 2012].
* Dyspnoea: A score of ≥1 on the Modified Medical Research Council Dyspnoea Scale (mMRC) at Visit 1.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known α-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease. Allergic rhinitis is not exclusionary.
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Exacerbations: Has had more than 1 moderate or severe COPD exacerbation in the past 12 months. Subjects with a moderate exacerbation within 6 weeks or severe exacerbations within 10 weeks prior to Visit 1 are excluded from study.

A moderate COPD exacerbation is defined as worsening symptoms of COPD that require treatment with oral/systemic corticosteroids and/or antibiotics. A severe exacerbation is defined as worsening symptoms of COPD that require in-patient hospitalization.

* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
* 12-Lead ECG: An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1, including the presence of a paced rhythm on a 12-lead ECG which causes the underlying rhythm and ECG to be obscured. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. Specific ECG findings that preclude subject eligibility are listed in Appendix 3. The study investigator will determine the medical significance of any ECG abnormalities not listed in Appendix 3.

Appendix 3:

* Sinus tachycardia ≥120 bpm. *Note: sinus tachycardia ≥120bpm should be confirmed by two additional readings at least 5 minutes apart.
* Sinus bradycardia <45bpm. *Note: Sinus bradycardia <45bpm should be confirmed by two additional readings at least 5 minutes apart.
* Multifocal atrial tachycardia.
* Supraventricular tachycardia (>100bpm).
* Atrial fibrillation with rapid ventricular response (rate >120bpm).
* Atrial flutter with rapid ventricular response (rate >120bpm).
* Ventricular tachycardias (non sustained, sustained, polymorphic, or monomorphic).
* Ventricular flutter.
* Ventricular fibrillation.
* Torsades de Pointes.
* Evidence of Mobitz type II second degree or third degree atrioventricular (AV) block.
* AV dissociation.
* 2:1 AV block.
* Trifascicular Block.
* For subjects with QRS duration <120 ms: QTc(F) ≥450msec or an ECG that is unsuitable for QT measurements (e.g., poor defined termination of the T wave).
* For subjects with QRS duration≥120: QTc(F) ≥480msec or an ECG that is unsuitable for QT measurements (e.g., poor defined termination of the T wave).
* Myocardial infarction (acute or recent) * Note: Evidence of an old (resolved) myocardial infarction is not exclusionary

  * Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
  * Medications Prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1.

Use as maintenance treatment in the 3 months prior to Visit 1 is not permitted. Maintenance treatment is defined as use for ≥ 14 consecutive days (at any time in the 3 months prior to Visit 1).

* Inhaled Corticosteroid (ICS)/Inhaled long acting beta2-agonists combinations
* Phosphodiesterase 4 (PDE4) inhibitors
* LABA
* Other Long acting muscarinic antagonists (does not include tiotropium)
* LAMA/LABA combinations
* Theophyllines
* Oral beta2-agonists (long-acting and short-acting) Use within 12 weeks is not permitted.
* Depot corticosteroids Use within 6 weeks is not permitted.
* Systemic, oral or parenteral corticosteroids
* Antibiotics (for lower respiratory tract infection)
* Cytochrome P450 3A4 strong inhibitors Use within 4 hours is not permitted.
* Inhaled short acting beta2-agonists, short-acting anticholinergics, and short-acting anticholinergic/short- acting beta2-agonist combination products (Use of study provided prn albuterol/salbutamol is permitted during the study, except in the 4-hour period prior to spirometry testing. Subjects who are taking short acting bronchodilators (beta-agonists or muscarinic antagonists) as their only form of bronchodilation at screening may NOT be recruited into the study).

Any other investigational medication use within 30 days or within 5 drug half-lives (whichever is longer) is not permitted

Note: if a LABA, LAMA (non-tiotropium), ICS/LABA, LAMA/LABA, theophylline, oral beta-agonist,or PDE4 inhibitor was taken on a non-maintenance basis (i.e., < 14 consecutive days over the 3 months prior to screening) the following minimum washouts must be observed prior to visit 1: twice-daily LABAs and ICS/LABAs = 48 hours; once-daily LABAs and ICS/LABAs= 14 days; LAMAs (excluding tiotropium) = 7 days; once-daily LAMA/LABA = 14 days, twice-daily LAMA/LABA = 7days; theophyllines = 48 hours; oral beta2 agonists = 48 hours; PDE4 inhibitor = 14 days.

* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., ≤12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 12 weeks prior to Visit 1 or are in the maintenance phase of a pulmonary rehabilitation program are excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Inability to Read: In the opinion of the investigator, any subject who is unable to read and/or write would not be able to complete a questionnaire.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2015-07-22 (Actual); Study Completion 2015-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (3):
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
- Argentina (5):
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (7):
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
- Norway (6):
  - GSK Investigational Site, Bodø
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Haugesund
  - GSK Investigational Site, Kløfta
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Tønsberg
- Russia (7):
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
- South Africa (7):
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Middelburg
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Somerset West
- GSK Investigational Site, Gyeonggi-do, South Korea
- Sweden (6):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Luleå
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
- Ukraine (5):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolayiv
  - GSK Investigational Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 116960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants (par) completed a 4-week open label tiotropium run-in phase, and were randomized to blinded study medication for 12 weeks. Supplemental albuterol/salbutamol was provided to all par, to be used on an as-needed basis during the run-in phase and up to Day 85.
Pre-assignment Details: A total of 739 par were enrolled; 496 par randomized and 494 par were included in the Intent-to-Treat (ITT) Population (Pop), comprised of all par randomized to treatment (trt) who received at least 1 dose of randomized study medication in the trt period.
Groups:
- Umeclidinium/Vilanterol 62.5/25 µg: Participants self-administered one dose of umeclidinium/vilanterol inhalation powder 62.5/25 micrograms (µg) once daily via an ELLIPTA dry powder inhaler and placebo once daily via a HANDIHALER each morning for 12 weeks. Each inhaler containing placebo was identical in appearance to its corresponding inhaler containing active study medication.
- Tiotropium Bromide 18 µg: Participants self-administered one dose of tiotropium bromide 18 µg once daily via a HANDIHALER and placebo once daily via an ELLIPTA dry powder inhaler each morning for 12 weeks. Each inhaler containing placebo was identical in appearance to its corresponding inhaler containing active study medication.
Period: Overall Study
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Tiotropium Bromide 18 µg
Started | 247 | 247
Completed | 230 | 231
Not Completed | 17 | 16
Not completed — Adverse Event | 5 | 4
Not completed — Lack of Efficacy | 1 | 5
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Umeclidinium/Vilanterol 62.5/25 µg: Participants self-administered one dose of umeclidinium/vilanterol inhalation powder 62.5/25 µg once daily via an ELLIPTA dry powder inhaler and placebo once daily via a HANDIHALER each morning for 12 weeks. Each inhaler containing placebo was identical in appearance to its corresponding inhaler containing active study medication.
- Total: Total of all reporting groups
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Tiotropium Bromide 18 µg | Total
Number analyzed (Participants) | 247 | 247 | 494
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (8.71) | 64.3 (8.74) | 64.4 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 87 | 171
  Male | 163 | 160 | 323
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 2 | 4 | 6
  Asian - Central/South Asian Heritage | 1 | 1 | 2
  White - Arabic/North African Heritage | 4 | 4 | 8
  White - White/Caucasian/European Heritage | 239 | 237 | 476
  White - Mixed Race | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) on Day 85 (Visit 8)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in 1 second. BL was the mean of the values measured 23 hour and 24 hour after dosing prior to Day 1 (ie. after the last open label [OL] tiotropium dosing and prior to the randomized dose). Change from BL is defined as the post-BL value minus the BL value. Trough FEV1 on Day 85 is defined as the mean of the FEV1 values obtained at 23 and 24 hours after dosing on Day 84 (at Week 12 + 1 day). Analysis performed using a mixed repeated measures model (MMRM) with covariates of treatment, BL, center group, 24 hour subset flag, Day, Day by BL and Day by treatment interactions. ITT Population is defined as participants who received at least one dose of randomized study medication in the treatment period. Only those participants with data available at the specified time point were included in the analysis.
Time Frame: Baseline (BL) and Day 85
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Tiotropium Bromide 18 µg
Number analyzed (Participants) | 224 | 225
Liters | 0.074 (0.0155) | -0.014 (0.0155)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol 62.5/25 µg vs Tiotropium Bromide 18 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.088, 95% CI 2-sided [0.045 to 0.131]

2. Secondary Outcome: Change From BL in FEV1 at 3 Hours Postdose on Day 84
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in 1 second. FEV1 assessments taken on 0 to 3 hour on Day 84 (pre-dose, 5 minutes (min), 15 min, 30 min, 1 hour, and 3 hour post-dose). Pre-dose was the reading obtained at 24 hours after the previous day's dose (Day 83 dose). BL is defined as mean of the values measured 23 hour and 24 hour after dosing prior to Day 1 (ie. after the last OL tiotropium dosing and prior to the randomized dose). Change from BL is defined as the post-BL value minus the BL value. Analysis performed using mixed model repeated measures with covariates of treatment, BL FEV1, center group, 24 hour subset flag, time, time by treatment interaction and time by BL interaction. Only those participants with data available at the specified time point were included in the analysis.
Time Frame: Baseline and Day 84
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Tiotropium Bromide 18 µg
Number analyzed (Participants) | 225 | 228
Liters | 0.164 (0.0178) | 0.091 (0.0177)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol 62.5/25 µg vs Tiotropium Bromide 18 µg; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 0.073, 95% CI 2-sided [0.024 to 0.122]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected over a period of a maximum of 94 days starting from Day 1 of treatment until the follow-up contact.
Description: On-treatment SAEs and non-serious AEs were reported for members of the ITT Population, comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Tiotropium Bromide 18 µg
Serious Adverse Events (participants affected / at risk) | 7/247 | 6/247
Other Adverse Events (participants affected / at risk) | 34/247 | 34/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Umeclidinium/Vilanterol 62.5/25 µg (N=247) | Tiotropium Bromide 18 µg (N=247)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Umeclidinium/Vilanterol 62.5/25 µg (N=247) | Tiotropium Bromide 18 µg (N=247)
Nasopharyngitis (Infections and infestations) | 18 | 17
Headache (Nervous system disorders) | 16 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.